CLINICAL TRIAL: NCT05537350
Title: A 12 Weeks of Clinical Study to Evaluate the Efficacy and Consumer Perception of Different Skin Attributes Following Supplementation of an Oral Supplement- Lumenato
Brief Title: A Clinical Study to Evaluate the Efficacy and Consumer Perception of Lumenato
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LycoRed Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CRLNJ2021-0990 BI
Record Dates: First submitted 2022-05-11; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Skin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumenato (Experimental): 1 Lumenato soft gel once a day
  Interventions: Dietary Supplement: Lumenato
- Placebo (Placebo Comparator): 1 Soft gels without active ingredients once a day
  Interventions: Dietary Supplement: Lumenato

INTERVENTIONS:
Dietary Supplement: Lumenato — Supplementation of 12 weeks

SUMMARY:
Subjects will be enrolled in this clinical study to assess the efficacy of an oral supplement to change the characteristics of facial skin after 4 and 12 weeks of use and obtain consumer perception of the test product through the use of questionnaires.

Study evaluations will include a comprehensive metabolic panel, Cutometer measurements, Canfield's VISIA-CR images, VapoMeter Measurements, and Consumer perception questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is female between 35 and 55 years of age;
2. Subject has a Fitzpatrick skin type of II, III, or IV;
3. Subject is of Caucasian or Latino;
4. Subject has self-perceived sensitive skin (defined as being sensitive to different topical products through different seasons resulting in any of the following: redness, irritation, itching, tingling, or edema);
5. Subject to have a baseline TEWL of ≥12;
6. Subject to have Glogau skin classification of Type 2 (see Appendix IV);
7. Subject is willing to get their blood drawn at Baseline and Week 4;
8. Subject is not currently enrolled in, and agrees not to participate in, any other oral nutritional supplement or face studies while enrolled in this study;
9. Subject agrees not to introduce any new nutricosmetic, cosmetic or toiletry products during the study;
10. Subject is dependable and able to follow directions as outlined in the protocol and anticipates being available for all study visits;
11. Subject is willing to participate in all study evaluations;
12. Subject is in generally good health and has a current Panelist Profile Form on file at CRL;
13. Subject agrees to sign a Photography Release Form, providing consent for the capture of digital images for use in relation to this clinical study ;
14. Subject has completed a HIPAA Authorization Form in conformance with 45 CFR Parts 160 and 164;
15. Subject understands and is willing to sign an Informed Consent Form in conformance with 21 CFR Part 50: "Protection of Human Subjects."

Exclusion Criteria:

1. Subject is pregnant, nursing, planning a pregnancy, or not using adequate birth control;
2. Subject has a history of digestive problems;
3. Subject is on blood thinners;
4. Subject has received treatment with sympathomimetics, antihistamines, vasoconstrictors, non-steroidal anti-inflammatory agents, and/or systemic or topical corticosteroids within 4 week prior to initiation of the study;
5. Chronic or relapsing inflammatory and/or allergic skin conditions such as atopic dermatitis, rosacea, psoriasis and alike including telangiectasias ("spider veins");
6. Current diagnosis of adult acne or currently on treatment for adult acne;
7. Participants who have received facial irradiation within last year or are planning on undergoing facial irradiation during the study;
8. Participants who currently take supplements containing carotenoids, lutein, melatonin or tryptophan;
9. Participants who use tanning salons or tanning products in the last 3 months;
10. Participants who plan to undergo invasive facial procedures (injections, chemical peeling, etc.) during the study or have undergone these procedures within 2 months prior to enrollment;
11. Participants with auto-immune skin diseases (e.g. scleroderma, psoriasis, lupus, epidermolysis bullosa, bullous pemphigoid, temporal arteritis);
12. Participants who have been prescribed retinoids treatment (<2 months prior to enrollment);
13. Current smokers;
14. Subject has a history of acute or chronic dermatologic, medical, and/or physical conditions which would, in the opinion of the Principal Investigator, preclude application of the test material and/or could influence the outcome of the study;
15. Subject is currently taking certain medications which, in the opinion of the Principal Investigator, may interfere with the study;
16. Subject is not willing to participate in all study evaluations;
17. Subject has known allergies to skin treatment products or cosmetics, toiletries, nutraceuticals, nutricosmetic, and/or topical drugs;
18. Subject has a history of skin cancer, or is currently undergoing treatment for active cancer of any kind;
19. Subject has diabetes.

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Improvment of skin barier as mesured by VapoMeter and FaceQ questionnaire | 12 weeks of use
  VapoMeter Measurements before and after treatment FaceQ questionnaire before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofins | CRL, Inc., Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No